CLINICAL TRIAL: NCT06354972
Title: Impact of the Senescence Associated Secretory Phenotype in the Gingival Crevicular Fluid on the Outcomes of Periodontal Regeneration
Brief Title: Impact of SASP in the GCF on the Outcomes of Periodontal Regeneration
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: SASP Turin
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minimally invasive periodontal regeneration: Minimally-invasive surgical technique (MIST) procedure using both biological inductors and bone xenograft.
  Interventions: Procedure: Minimally invasive surgical procedure

INTERVENTIONS:
Procedure: Minimally invasive surgical procedure — All the experimental sites underwent a minimally-invasive surgical technique (MIST) procedure under magnification (Cortellini and Tonetti 2007). The full-thickness flap was minimally raised both on the buccal and oral side, avoiding vertical releasing incisions. Granulation tissue was scraped from the bony surfaces of the defect, and the root was debrided using minicurettes/ultrasonic device and chemically treated by EDTA. Regenerative procedure was carried out using a combination of enamel matrix derivatives and bone xenograft. The flaps were then repositioned and sutured in order to obtain passive primary closure.

SUMMARY:
Objectives: To test the impact of clinical inflammation and molecular expression profile (senescence-associated secretory phenotype; SASP) in the gingival crevicular fluid (GCF) on the outcomes of minimally-invasive periodontal regeneration in intra-bony defects.

Methods: Sites associated with intrabony defects ≥ 3 mm requiring periodontal regeneration through minimally-invasive surgical technique were included. Pre-operatively, GCF was sampled for inflammatory biomarker analysis related to SASP [interleukin (IL)-1β, IL-6 and IL-12; matrix-metalloproteinases (MMP)-8 and -9]. Correlation analyses and logistic regression models were performed to assess the impact of predictors on clinical and radiographic outcomes.

ELIGIBILITY:
Inclusion criteria comprised:

1) diagnosis of stage III or IV periodontitis (Papapanou et al. 2018b); 2) full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) of <15%; 3) completion of steps I-II of periodontal treatment at least 2 months priorly; 4) tooth with residual PPD ≥ 6 mm, BoP+, and a radiographic intrabony component ≥ 3 mm, lacking furcation involvement (Aimetti et al. 2023), considered suitable for a minimally invasive procedure (Cortellini and Tonetti 2007) (Fig. 1A).

Exclusion criteria encompassed:

1) age < 18 years; 2) current smokers; 3) contraindications to surgery; 4) systemic diseases that could impact periodontal healing; 5) pregnancy and lactation; 6) a history of periodontal surgery at the experimental teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a diagnosis of stage III or IV periodontitis who had undergone steps I-II of periodontal therapy were considered for inclusion.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change | [Time Frame: 12 months]
  Clinical attachment level will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Achievement of composite outcome measure | [Time Frame: 12 months]
  Composite outcome measure (COM) will be achieved by sites with probing pocket depth < 4 mm and relevant clinical attachment gain ≥ 3 mm at the 12-month re-evaluation

SECONDARY OUTCOMES:
Radiographic bone level change | [Time Frame: 12 months]
  Periapical standardized radiographs will be taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)
Probing pocket depth change | [Time Frame: 12 months]
  Probing depth will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: No